CLINICAL TRIAL: NCT02490449
Title: Dexlansoprazole MR in Nonerosive Reflux Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Su Jin Hong, professor, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBC 2014-05-021-002
Record Dates: First submitted 2014-12-13; First posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Nonerosive Reflux Disease

ARMS (2):
- Exprerimental group (Experimental): medication after diet
  Interventions: Drug: Dexlansoprazole MR
- control group (Active Comparator): medication before diet
  Interventions: Drug: Dexlansoprazole MR

INTERVENTIONS:
Drug: Dexlansoprazole MR — Administration of drug after or before diet

SUMMARY:
This study aim is to compare the efficacy of Dexlansoprazole MR intake before and after breakfast in patients with nonerosive reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* NERD confirmed by gastroscopy

Exclusion Criteria:

* PPI medication within 2 weeks before enrollment

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Percentage (%) of patients free of reflux symptoms | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Su Jin Hong, Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Digestive Disease Center, Department of Internal Medicine, Soonchunhyang University College of Medicine, Bucheon-si, Gyeonggi-do, South Korea